CLINICAL TRIAL: NCT01824394
Title: reMARQable nMARQ™ Pulmonary Vein Isolation System for the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: nMARQ™ Pulmonary Vein Isolation System for the Treatment of Paroxysmal Atrial Fibrillation
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: reMARQable
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: nMARQ; Atrial Fibrillation; Drug Refractory; Radio Frequency
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- nMARQ Catheter (Experimental): nMARQ Catheter System
  Interventions: Device: nMARQ Navigation Catheters
- NaviStar ThermoCool Catheters (Active Comparator): THERMOCOOL® Navigational family of catheters
  Interventions: Device: NaviStar ThermoCool Catheters

INTERVENTIONS:
Device: nMARQ Navigation Catheters
  Arms: nMARQ Catheter
Device: NaviStar ThermoCool Catheters
  Arms: NaviStar ThermoCool Catheters

SUMMARY:
To demonstrate safety and effectiveness of nMARQ Catheter System [nMARQ] compared with THERMOCOOL® Navigational Family of catheters in treating subjects with drug-refractory symptomatic paroxysmal atrial fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic paroxysmal AF who have had at least one AF episode documented within one (1) year prior to enrollment. Documentation may include ECG, transtelephonic monitor (TTM), Holter monitor (HM), or telemetry strip.
2. Patients who have failed at least one antiarrhythmic drug (AAD; class I or III, or atrioventricular (AV) nodal blocking agents such as beta blockers and calcium channel blockers) as evidenced by recurrent symptomatic AF, or intolerance to the AAD.
3. Pre-procedure anticoagulation on warfarin, rivaroxaban, or apixaban.
4. Age 18 years or older.
5. Signed Patient Informed Consent Form (ICF).
6. Able and willing to comply with all pre-, post-, and follow-up testing and requirements.

Exclusion Criteria:

1. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
2. Previous ablation for atrial fibrillation.
3. Patients on amiodarone at any time during the past 3 months prior to enrollment.
4. AF episodes lasting > 7 days.
5. Any cardiac surgery within the past 60 days (2 months).
6. Any valvular cardiac surgical procedure (i.e., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve).
7. Coronary artery bypass graft (CABG) procedure within the last 180 days (6 months).
8. Awaiting cardiac transplantation or other cardiac surgery within the next 365 days (12 months).
9. Documented left atrial thrombus on imaging.
10. History of a documented thromboembolic event within the past one (1) year.
11. Diagnosed atrial myxoma.
12. Presence of implanted cardioverter defibrillator (ICD).
13. Significant pulmonary disease, (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
14. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
15. Women who are pregnant (as evidenced by pregnancy test if subject is of child-bearing age and potential) or breast feeding.
16. Acute illness or active systemic infection or sepsis.
17. Unstable angina.
18. Myocardial infarction within the previous 60 days (2 months).
19. Left ventricular ejection fraction <40%.
20. History of blood clotting or bleeding abnormalities.
21. Contraindication to anticoagulation (i.e., heparin, dabigatran, Vitamin K Antagonists such as warfarin).
22. Life expectancy less than 365 days (12 months).
23. Enrollment in an investigational study evaluating another device or drug.
24. Uncontrolled heart failure or NYHA Class III or IV heart failure.
25. Presence of intramural thrombus, tumor or other abnormality that precludes catheter introduction or manipulation.
26. Presence of a condition that precludes vascular access.
27. Left atrial size >50 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2017-11-26 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on April 1, 2013. Enrollment was terminated on May 25, 2017.
Pre-assignment Details: This was a prospective, multicenter, randomized, controlled, two arm single-blind design. Enrolled subjects N=481 (subjects signed informed consent) 468 does not include 13 subjects excluded prior to randomization.
Groups:
- nMARQ® Group: Pulmonary vein isolation by radiofrequency ablation treatment with the nMARQ® catheter.
- ThermoCool Group: Pulmonary vein isolation by radiofrequency ablation treatment with the THERMOCOOL® catheter.
- Roll-in Subjects: Calibration roll-in cohort
Period: Overall Study
Arm/Group | nMARQ® Group | ThermoCool Group | Roll-in Subjects
Started (Patients who signed informed consent forms) | 174 | 169 | 125
Intent to Treat Population (Intent-to-Treat (ITT) population include randomized patients who have the ablation catheter inserted) | 151 | 149 | 0 (Calibration Roll-in patients are not included in the ITT)
Safety Population (Safety Population includes those patients who have the ablation catheter inserted) | 151 | 149 | 104 (Calibration Roll-in patients are included in the safety population)
Per-Protocol Population (Includes ITT patients who have undergone RF ablation and are in compliance with study protocol) | 150 | 148 | 0 (Calibration Roll-in patients are not included in the per protocol population)
Completed (All enrolled subjects who underwent insertion of the study catheter) | 55 | 53 | 51
Not Completed | 119 | 116 | 74
Not completed — Early Termination | 1 | 1 | 3
Not completed — Withdrawn due to Study Termination | 91 | 83 | 41
Not completed — Lost to Follow-up | 0 | 9 | 3
Not completed — Death | 3 | 2 | 4
Not completed — Discontinued Subjects | 1 | 1 | 2
Not completed — Excluded Subjects(No catheter inserted) | 23 | 20 | 21

BASELINE CHARACTERISTICS:
Population: Enrolled subjects N=481 (subjects signed informed consent) 468 does not include 13 subjects; 10 subjects excluded prior to randomization, 3 excluded subjects missing data.
Groups:
- THERMOCOOL® Group: Pulmonary vein isolation by radiofrequency ablation treatment with the THERMOCOOL® catheter.
- Total: Total of all reporting groups
Arm/Group | nMARQ® Group | THERMOCOOL® Group | Roll-in Subjects | Total
Number analyzed (Participants) | 174 | 169 | 125 | 468
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Only include those enrolled subjects with data available. Enrolled subjects are those who signed informed consent forms.
  Years | 62.0 (10.81) | 61.8 (10.40) | 63.6 (9.96) | 62.4 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Enrolled subjects with data available.
  Participants
    Female | 66 | 60 | 50 | 176
    Male | 108 | 109 | 75 | 292
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Enrolled Subjects with data available. 467 does not include 14 subjects; 1 ThermoCool group patient missing data, 9 subjects excluded prior to randomization, 4 excluded subjects missing data.
  Participants
    number analyzed (Participants) | 174 | 168 | 125 | 467
    Hispanic or Latino | 6 | 3 | 5 | 14
    Not Hispanic or Latino | 168 | 165 | 120 | 453
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Enrolled subjects with data available.
  Participants
    American Indian or Alaska Native | 0 | 2 | 1 | 3
    Asian | 2 | 0 | 1 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 2 | 0 | 0 | 2
    White | 169 | 165 | 121 | 455
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Early Onset Primary Adverse Events
Description: The primary safety endpoint was the incidence of early-onset primary adverse events within 7 days post the AF ablation procedure; Pulmonary vein stenosis and atrio-esophageal fistula that occurred beyond 7 days post-procedure and development of a significant pericardial effusion within 30 days post-procedure were also considered primary AEs
Time Frame: 30 days post-procedure
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | nMARQ® Group | ThermoCool Group | Roll-in Subjects
Number analyzed (Participants) | 151 | 149 | 104
Participants | 8 | 7 | 9

2. Primary Outcome: Incidence of Early Onset Primary Adverse Events for the Intent-to-Treat and As-Treated Population
Description: as for outcome 1
Time Frame: 30 days post-procedure
Population: The Intent-to-Treat and As-Treated population which includes randomized patients who have the ablation catheter inserted
Measure: Count of Participants; unit: Participants
Arm/Group | nMARQ® Group | ThermoCool Group
Number analyzed (Participants) | 151 | 149
Participants | 8 | 7

ADVERSE EVENTS:
Time Frame: 3 years post ablation procedures
Arm/Group | nMARQ® Group | THERMOCOOL® Group | Roll-in Subjects
All-Cause Mortality (participants affected / at risk) | 3/151 | 2/149 | 4/104
Serious Adverse Events (participants affected / at risk) | 38/151 | 25/149 | 31/104
Other Adverse Events (participants affected / at risk) | 86/151 | 86/149 | 74/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nMARQ® Group (N=151) | THERMOCOOL® Group (N=149) | Roll-in Subjects (N=104)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ependymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic lymphocytic leukaemia (in remission) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 4 (5)
Atrial flutter (Cardiac disorders) | 6 (11) | 2 (2) | 2 (3)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Cardiac disorders) | 0 (0) | 1 (1) | 4 (4)
Fluid overload (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Pericardial effusion (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2)
Presyncope (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (3) | 1 (1)
Goitre (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocele (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal cancer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 1 (2)
Device related infection (General disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Phrenic nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Explorative laparotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Meniscus operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Oesophagogastric fundoplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Vascular pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nMARQ® Group (N=151) | THERMOCOOL® Group (N=149) | Roll-in Subjects (N=104)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (6) | 3 (3) | 4 (8)
Bradycardia (Cardiac disorders) | 4 (4) | 1 (1) | 2 (2)
Chest pain (Cardiac disorders) | 1 (10) | 1 (11) | 6 (9)
Dyspnoea (Cardiac disorders) | 3 (3) | 2 (2) | 2 (2)
Fluid overload (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2)
Oedema peripheral (Cardiac disorders) | 2 (3) | 2 (3) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Pericardial effusion (Cardiac disorders) | 6 (6) | 4 (4) | 7 (7)
Presyncope (Cardiac disorders) | 2 (2) | 2 (2) | 4 (4)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Syncope (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 5 (5) | 4 (4) | 5 (6)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Thyroid disorder (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Corneal abrasionCorneal abrasion (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Oesophageal injury (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (3) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 4 (4) | 1 (1)
Vessel puncture site haematoma (General disorders) | 1 (1) | 1 (1) | 3 (3)
Hypersensitivity (Immune system disorders) | 5 (5) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4) | 0 (0) | 4 (5)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 3 (4) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 1 (1) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (10) | 1 (1) | 4 (4)
Heart rate increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 1 (1)
Dysphonia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Sleep apnoea syndrome (Nervous system disorders) | 5 (5) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Haematuria (Renal and urinary disorders) | 4 (4) | 2 (2) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (11) | 7 (7) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 9 (10) | 8 (9) | 7 (8)
Hypotension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for 60 to 180 days from the time submitted to the sponsor for review. For multicenter studies, the first results communications should be a joint multicenter publication. PIs may communicate results from their institution as indicated above if a multicenter publication is not submitted by the Sponsor or representatives within 12 months of the study's conclusion.

DOCUMENTS (2):
  • Study Protocol (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT01824394/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT01824394/SAP_001.pdf